CLINICAL TRIAL: NCT07013227
Title: The Effect of Virtual Reality Glasses Application on Labor Pain and Comfort in Multiparous Pregnants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Çiğdem, Assistant Proffesor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: MarmaraUEbelik
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Labor Pain
Keywords: birth; labor pain; virtual reality glasses
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): It refers to the group in which virtual reality glasses will not be applied.
- experimental group (Experimental): It refers to the group to which virtual reality glasses will be applied.
  Interventions: Other: experimental group

INTERVENTIONS:
Other: experimental group — Labor pain and comfort level will be measured by applying virtual reality glasses to the control group.
  Arms: experimental group

SUMMARY:
One of the non-pharmacological methods used to reduce labor pain in multiparous pregnant women is the application of virtual reality glasses. This study aims to measure labor pain and determine the effect of virtual reality glasses application on comfort.

DETAILED DESCRIPTION:
One of the non-pharmacological methods in the management, control and reduction of labor pain is the application of virtual reality glasses. Non-pharmacological methods applied by midwives in obstetrics clinics are preferred because they do not have any side effects to the mother and fetus, their cost is very low and they are easy to apply.

This study was planned to determine the effect of virtual reality glasses application on labor pain and comfort in multiparous pregnant women.

The research was planned at Istanbul Sultanbeyli State Hospital between 15 September 2023 and 31 June 2024. The universe of the research will be the pregnant women who were hospitalized to give birth in this hospital, and the sample will be multiparous pregnant women (60 experimental group, 60 control group) who are in the active phase of labor and comply with the sampling criteria, and a total of 120 pregnant women. Block randomization will be used in sample selection. Those who volunteered to participate in the study will have to sign the Informed Consent Form, and the Pregnant Woman Descriptive Information Form, Visual analog scale-VAS, Comfort Scale-QL and Birth Satisfaction Scale will be filled in by the researchers by face-to-face interview technique. Data collection will take approximately 15-20 minutes.As a result of the study, to reveal the effectiveness of virtual reality glasses application, which is one of the non-pharmacological methods, in reducing labor pain and increasing the birth comfort and satisfaction of mothers, and to contribute to the literature in this field by adding a new one to the limited studies in this field. This study was planned as a randomized controlled experimental study to determine the effect of virtual reality glasses application on labor pain and comfort in multiparous pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-35
* At least primary school graduate
* Able to speak and understand Turkish
* 37-42 weeks of pregnancy (term)
* Having a singleton pregnancy
* Fetal presentation is head
* Vaginal birth planned
* Multiparity (2 or more births)
* Does not have any risks related to pregnancy and birth
* There is no problem in the fetus
* In the active phase of labor
* Pregnant women who volunteer to participate in the study and approve the consent document will be included.

Exclusion Criteria:

* Those under the age of 18 (Adolescents)
* Primiparity (First to give birth)
* Those who are planned to have a caesarean section
* Analgesics administered at birth
* Those who did not want to participate in the study or participated in the study voluntarily but later those who give up

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
birth comfort scale | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: zümrüt bilgin, Study Director — Marmara University
Locations (1):
- Marmara University Faculty of Health Sciences, Istanbul, Turkey (Türkiye)